CLINICAL TRIAL: NCT02917434
Title: Effects of Weight-loss Treatment in Obese Patients With Psoriatic Arthritis
Acronym: VIPsA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 211861
Record Dates: First submitted 2016-09-21; First posted 2016-09-28 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2020-05

CONDITIONS: Obesity; Psoriatic Arthritis; Metabolic Syndrome; Psoriasis; Cardiovascular Disease
Keywords: Obesity; Psoriatic arthritis; Psoriasis; Metabolic syndrome; Cardiovascular disease
MeSH Terms: conditions — Obesity; Arthritis, Psoriatic; Metabolic Syndrome; Psoriasis; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with PsA and obesity (Active Comparator): Very Low Energy Diet (VLED)
  Interventions: Dietary Supplement: Very Low Energy Diet (VLED)
- Patients with obesity (Other): Very Low Energy Diet (VLED)
  Interventions: Dietary Supplement: Very Low Energy Diet (VLED)

INTERVENTIONS:
Dietary Supplement: Very Low Energy Diet (VLED) — Very Low Energy Diet (VLED), divided into 4 daily doses, gives any intake of 640 calories per day together with the recommended doses of vitamins and minerals. During an initial period of 12 weeks the patients only consume VLED. After the strict period food is successively reintroduced during a period of 18 weeks.

SUMMARY:
The study is an open intervention study with the aim to determine the effects of weight-loss treatment with Low-Energy liquid Diet (LED) on disease activity, quality of life and markers of the metabolic syndrome in patients with psoriatic arthritis and obesity.

DETAILED DESCRIPTION:
BACKGROUND Psoriasis is a common skin disease affecting around 2-3% of the population in Sweden. Approximately 20-30% of the individuals with psoriasis develop psoriatic arthritis (PsA). PsA mainly engage the musculoskeletal apparatus and causes inflammation of joints, tendons and ligaments, but the disease also increases the risk of developing anterior uveitis and inflammatory bowel disease, especially Crohn's disease.

Both psoriasis and PsA are strongly associated with obesity and the metabolic syndrome (Mets). Observational studies have reported a frequency of obesity (body mass index; BMI≥30 kg/m2) in 45% and of MetS in 30-45% of PsA patients. Earlier studies have shown that obesity increases the risk of developing both psoriasis and PsA and that obesity is associated with increased disease activity, poorer treatment response and lower chance of achieving minimal disease activity.

Although the association between PsA and obesity is well known, there are only a small number of interventional studies which have assessed the effects of weight loss on disease activity in PsA.

Patients with PsA also have an increased risk of cardiovascular disease. [12, 13] Chronic inflammation, which accelerates the atherosclerotic process, in combination with a higher prevalence of cardiovascular risk factors among PsA patients is believed to contribute to this increased risk.

Obesity causes a low grade systemic inflammation via the production of pro-inflammatory mediators in the white adipose tissue, such as adipokines and cytokines (e.g. tumour necrosis factor-α and interleukin-6), which are also involved in the pathogenic process if PsA. Obesity-related inflammation could thus act synergistically with autoimmune inflammation in the development and the maintenance of disease in psoriasis and PsA.

Weight-loss treatment with Very Low Energy Diet (VLED) is an effective and approved method in clinical use in Sweden. In severe obesity, BMI 35 kg/m2 or more, a strict energy restriction is needed for optimal weight-loss. The LED gives a daily intake of 640 calories together with the recommended doses of vitamins and minerals. During an initial period of 12 weeks the patients only consume LED. The weight-loss with this intake is 1-2 kilograms per weeks. After the strict period food is successively reintroduced during a period of 18 weeks. The treatment is given within the framework of a structured program including support and medical follow-up from a team of doctors, nurses and dieticians.

AIMS The aims of this study are

* To determine the effects of weight loss treatment on disease activity, function, quality of life and markers for the metabolic syndrome in patients with psoriatic arthritis
* To study the specific effects on the immune system of the negative energy balance during the strict energy restriction period and prospectively, during a two year follow-up
* To investigate if there are differences in body-composition, markers for Mets and adipokines between patients with PsA and obesity and controls with obesity before during and after weight loss treatment.

PATIENTS AND METHODS Patients with PsA and obesity registered at the Rheumatology clinics of Sahlgrenska University hospital and the hospitals of Alingsås and Borås are invited to participate.

The results of the PsA patients will be compared with control patients with obesity (PsA or psoriasis) matched for age, sex and BMI who undergo the same weight loss treatment with VLED.

Disease activity, physical function and quality of life will be assessed by physical examination (including anthropometric measures, joints, tendons, back mobility and skin) and by validated questionnaires at baseline (start of weight-loss treatment), 3 months, 6 months, 12 months and 24 months. Blood samples will be collected at the same appointments.

Body-composition will be measured at baseline and 12 months. Muscle strengths and physical function will be measured at baseline, 6 months and 12 months and physical activity will be assessed with questionnaires and accelerometers.

Informed written consent will be obtained from all patients and controls. The study was approved by the local regional ethics committee in Gothenburg and will be carried out in accordance with the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* PsA fulfilling the Classification for Psoriatic Arthritis (CASPAR) criteria
* BMI≥33 kg/m2
* Age 18-75 years

Exclusion Criteria:

* Pregnancy
* Porphyria
* Epilepsy
* Diabetes type 1
* Severe heart or kidney disease
* Eating disorder
* Severe catabolic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-04; Primary Completion 2019-12-12 (Actual); Study Completion 2021-10-06 (Actual)

PRIMARY OUTCOMES:
Minimal Disease Activity (MDA) which is a composite outcome measure | 6 months
  5 of 7 of the following criteria: Tender joint count ≤ 1 Swollen joint count ≤ 1 PASI ≤ 1or BSA ≤ 3 Patient pain VAS ≤ 15 Patient global activity VAS ≤ 20 HAQ ≤ 0.5 Tender entheseal points ≤ 1 BSA: body surface area; HAQ: Health Assessment Questionnaire; PASI

CONTACTS AND LOCATIONS:
Overall Officials: Eva Klingberg, M.D., Ph.D., Principal Investigator — Department of Rheumatology and Inflammation Research, Sahlgrenska Academy at the University of Gothenburg, Sweden
Locations (4):
- Sweden (4):
  - Department of Rheumatology at the Hospital of Alingsås, Alingsås
  - Department of Rheumatology at the Hospital of Borås, Borås
  - Department of Obesity and Internal Medicine at Sahlgrenska University Hospital, Gothenburg
  - Department of Rheumatology at Sahlgrenska University Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Torres L, Jonsson CA, Eliasson B, Forsblad-d'Elia H, Landgren AJ, Bilberg A, Gjertsson I, Larsson I, Klingberg E. A six-month weight loss intervention is associated with significant changes in serum biomarkers related to inflammation, bone and cartilage metabolism in obese patients with psoriatic arthritis and matched controls. BMC Rheumatol. 2025 May 23;9(1):58. doi: 10.1186/s41927-025-00511-0. PMID 40410839
- [Derived] Landgren AJ, Bilberg A, Eliasson B, Torres L, Dehlin M, Jacobsson LTH, Larsson I, Klingberg E. Health-related quality of life significantly improved in obese patients with psoriatic arthritis one year after a structured weight loss intervention. Adv Rheumatol. 2025 Mar 14;65(1):13. doi: 10.1186/s42358-025-00444-9. PMID 40087727
- [Derived] Landgren AJ, Jonsson CA, Bilberg A, Eliasson B, Torres L, Dehlin M, Jacobsson LTH, Gjertsson I, Larsson I, Klingberg E. Serum IL-23 significantly decreased in obese patients with psoriatic arthritis six months after a structured weight loss intervention. Arthritis Res Ther. 2023 Jul 27;25(1):131. doi: 10.1186/s13075-023-03105-8. PMID 37501212
- [Derived] Bilberg A, Larsson I, Bjorkman S, Eliasson B, Klingberg E. The impact of a structured weight-loss treatment on physical fitness in patients with psoriatic arthritis and obesity compared to matched controls: a prospective interventional study. Clin Rheumatol. 2022 Sep;41(9):2745-2754. doi: 10.1007/s10067-022-06164-5. Epub 2022 Jun 1. PMID 35648298
- [Derived] Klingberg E, Bjorkman S, Eliasson B, Larsson I, Bilberg A. Weight loss is associated with sustained improvement of disease activity and cardiovascular risk factors in patients with psoriatic arthritis and obesity: a prospective intervention study with two years of follow-up. Arthritis Res Ther. 2020 Oct 22;22(1):254. doi: 10.1186/s13075-020-02350-5. PMID 33092646
- [Derived] Klingberg E, Bilberg A, Bjorkman S, Hedberg M, Jacobsson L, Forsblad-d'Elia H, Carlsten H, Eliasson B, Larsson I. Weight loss improves disease activity in patients with psoriatic arthritis and obesity: an interventional study. Arthritis Res Ther. 2019 Jan 11;21(1):17. doi: 10.1186/s13075-019-1810-5. PMID 30635024